CLINICAL TRIAL: NCT04942548
Title: Reverse HFpEF: Ketogenic Reversal of Heart Failure With Preserved Ejection Fraction Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Darlene Kim, Associate Professor, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-3243 Keto
Record Dates: First submitted 2021-05-25; First posted 2021-06-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure
Keywords: obese; keto; diet; cardiac
MeSH Terms: conditions — Heart Failure; Obesity | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFpEF (Experimental): Patients diagnosed with obesity related heart failure with preserved ejection fraction(HFpEF)
  Interventions: Other: Ketogenic Diet
- PH-HFpEF (Experimental): Patients diagnosed with obesity related pulmonary hypertension heart failure with preserved ejection fraction (PH-HFpEF)
  Interventions: Other: Ketogenic Diet

INTERVENTIONS:
Other: Ketogenic Diet — Ketogenic diet intervention that is high in fat and low in carbohydrates, causing the body to induce a state of metabolic ketosis, whereby fat is broken down into ketones to provide an energy source for the body.

SUMMARY:
This protocol is a prospective pilot study utilizing the intervention of a medically supervised, registered nurse and registered diabetes educator coached low-carbohydrate, ketogenic diet to examine the impact it has as a treatment for heart failure with preserved ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 21-80) who meet clinical signs and symptoms of heart failure based on clinical assessment.
* The subject must meet at least one of the following hemodynamic criteria for HFpEF of PH-HFpEF by right heart catheterization (RHC) within 6 months of screening visit;

A) HFpEF:

1. At rest: mean pulmonary artery occlusions pressure (PAOP) > 15, pulmonary vascular resistance (PVR) < 3 Wood Units, or
2. HFpEF with fluid challenge, defined as increase in PAOP post 500 cc fluid bolus: mean PAOP > 18, PVR < 3 Wood Units, or
3. HFpEF with exercise, defined as peak mean PAOP > 17, PVR < 3 Wood Units if age < 50 or peak mean PAOP > 19 and PVR < 3 Wood Units if age >= 50

B) PH-HFpEF:

1. At rest: mean pulmonary artery occlusion pressure (PAOP) > 15, mean pulmonary artery pressure (PAP) >= 25, pulmonary vascular resistance (PVR) > 3 Wood Units, or
2. PH-HFpEF with fluid challenge, defined as increase in PAOP post 500 cc fluid bolus: mean PAOP > 18, mean PAP >= 25, PVR > 3 Wood Units, or
3. PH-HFpEF with exercise, defined as peak mean PAOP > 17, peak mean PAP > 30, peak PVR > 1.34 Wood Units if age < 50 or peak mean PAOP > 19, peak mean PAP > 33, and PVR < 2.1 Wood Units if age >= 50

   * The subject also must meet criteria for metabolic syndrome, defined as: Abdominal obesity (BMI > 30 kg/m2 or abdominal obesity, waist circumference > 102 cm men, > 88 cm women) AND 2 of the following;

a. Currently being treated for systemic hypertension or blood pressure (BP) >= 135/85 b. Glucose intolerance with diagnosis of type 2 diabetes, or fasting blood glucose 110-125 mg/dL or hemoglobin A1c > 6% c. Triglycerides >= 150, or on treatment for high triglycerides d. HDL < 40 men, < 50 women, or on treatment for high triglycerides

* If the subject is on pulmonary hypertension specific vasodilators, they must be on stable medical therapy without changes to pulmonary vasodilator medication within 3 months prior to screening visit.
* The subject must have also had a cardiopulmonary exercise test within 6 months of screening visit.
* The subject must have also had an echocardiogram within 6 months of screening visit.
* The subject must have demonstrated stable weight (less that 5% weight loss) 3 months prior to screening visit. (They cannot already be losing weight).
* The subject owns and uses a smartphone or tablet.
* Must speak English

Exclusion Criteria:

* The subject is already on a significant weight loss trajectory prior to study entry.
* The subject cannot be on an alternative diet plan or strategy (e.g., Weight Watchers, Nutrisystem, Ornish).
* Left ventricular ejection fraction < 50%.
* Severe valvular disease by echocardiogram or dysfunctional prosthetic valve.
* Active pericardial disease (moderate or large pericardial effusion or constrictive pericarditis).
* Active coronary ischemia defined by abnormal stress test, angiogram, or coronary CT angiography per investigator.
* Prolonged corrected QT interval (QTc) > 450 ms
* Significant lung disease on pulmonary function tests (PFT's) within the 6 months of screening visit, (Both post-bronchodilator values and pre-bronchodilator values must meet exclusion criteria. If either post- or pre-bronchodilator values do not, the subject may be included) defined as either:

  1. Irreversible obstructive airways disease (post-bronchodilator forced expiratory volume/forced vital capacity (FEV1/FVC) < 70% predicted) or
  2. Restrictive lung disease (FVC < 70% predicted. If total lung capacity (TLC) is >= 70%, it is acceptable to have an FVC of < 70%) or
  3. More than mild radiographic pulmonary disease as determine don CT scan within the past 2 years per investigator.
* History of non-adherence to diuretics within 3 months of screening visit.
* History or recurrent severe hypokalemia, potassium < 3.0 mg/dL.
* History of kidney stones, gout, or gallbladder disease unless in the opinion of the investigator it will not impact the safety of the patient
* C-peptide < 0.5 ng/mL (increased risk of diabetic ketoacidosis (DKA))
* Uncorrected anemia (hemoglobin < 10 g/dL).
* Unable to participate in the comprehensive ketogenic diet program, including biometric data acquisition and data entry (glucometer self-stick and smartphone use).
* Unable or unwilling to prepare meals for self.
* Unable to perform quantitative cardia testing regimen (cardiopulmonary exercise testing, 6-minute walk).
* Subject is pregnant or planning to become pregnant in the next 14 months.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
MLHFQ Questionnaire | 6 Months
  Change in score on the Minnesota Living with Heart Failure Quality of Life (MLHFQ) Questionnaire for the HFpEF cohort.
  * Max. Score = 105
  * Min. Score = 0
  * A reduced score means improvement of heart failure symptoms; better outcome
PAH-SYMPACT Questionnaire | 6 Months
  Change in score on the Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Questionnaire for the PH-HFpEF cohort.
  * Max. Score = 89
  * Min. Score = 0
  * A reduced score means improvement of pulmonary hypertension heart failure symptoms; better outcome

SECONDARY OUTCOMES:
Change in Metabolic Health: Weight | 6 Months
  Weight in kilograms (kg)
Change in Metabolic Health: Glucose | 6 Months
  Glucose in milligrams per deciliter (mg/dL)
Change in Metabolic Health: Insulin | 6 Months
  Insulin in microinternational unit per milliliter (uIU/mL)
Change in Metabolic Health: Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 6 Months
  Insulin and glucose are multiplied then divided by 405 to report HOMA-IR
Change in Metabolic Health: Albumin | 6 Months
  Albumin in grams per deciliter (g/dL)
Change in Metabolic Health: Bilirubin total | 6 Months
  Bilirubin total in milligrams per deciliter (mg/dL)
Change in Metabolic Health: Alanine Transaminase (ALT) | 6 Months
  ALT in units per liter (U/L)
Change in Metabolic Health: Aspartate Aminotransferase (AST) | 6 Months
  AST in units per liter (U/L)
Change in Metabolic Health: Alkaline Phosphatase (ALP) | 6 Months
  ALP in units per liter (U/L)
Change in Metabolic Health: High Sensitivity C-Reactive Protein (HS-CRP) | 6 Months
  HS-CRP in milligrams per deciliter (mg/dL)
Change in Metabolic Health: Triglycerides | 6 Months
  triglyceride in milligrams per deciliter (mg/dL)
Change in Metabolic Health: High Density Lipoprotein (HDL) | 6 Months
  HDL in milligrams per deciliter (mg/dL)
Change in Metabolic Health: Hemoglobin A1c | 6 Months
  hemoglobin A1c in percent (%)
Change in Metabolic Health: Body Mass Index (BMI) | 6 Months
  Weight and height will be combined to report BMI in kg/m^2
Changes in Physical Function: 6 Minute Walk Test (6MWT) | 6 Months
  6-minute walk test is reported in meters (m) of how far a subject walks in 6 minutes
Changes in Physical Function: Maximum Oxygen Consumption (VO2max) | 6 Months
  VO2 max is reported in liters per minute (L/min) while performing a cardiopulmonary exercise test (CPET)
Changes in Physical Function: Maximum Work | 6 Months
  Maximum work achieved while performing a cardiopulmonary exercise test (CPET) is reported in watts (W)
Changes in Physical Function: 30 Second Sit-to-Stand test (30s STS) | 6 Months
  30s STS is reported in quantity of how many times the subject can come to a full stand from a seated position in 30 seconds (s)
Changes in Physical Function: Leg Press - 1 Repetition Maximum | 6 Months
  Leg press is reported in kilograms (kg)
Changes in Physical Function: Chest Press - 1 Repetition Maximum | 6 Months
  Chest press is reported in kilograms (kg)
Changes in Physical Function: Leg Extension - 1 Repetition Maximum | 6 Months
  Leg extension is reported in kilograms (kg)
Cardiac Remodeling: Changes in the Left Ventricle (LV) size | 6 Months
  This is determined by the internal diameter measurement of the LV, reported in centimeters (cm) from a subject performed echocardiogram
Cardiac Remodeling: Changes in the Left Ventricle (LV) thickness | 6 Months
  This is determined by a measurement of the LV wall, reported in millimeters (mm) from an echocardiogram.
Cardiac Remodeling: Changes in the Left Ventricle (LV) mass | 6 Months
  This is determined by a combination formula of the interventricular septum diastole (IVSd), left ventricle diastole (LVd), and posterior wall diastole (PWd), calculated by an echocardiogram and reported in grams (g).
Cardiac Remodeling: Changes in Left Atrium (LA) size | 6 Months
  This is determined by the internal diameter measurement of the LA, reported in centimeters (cm) from a subject performed echocardiogram.
Cardiac Remodeling: Changes in Inferior Vena Cava (IVC) size | 6 Months
  This is determined by the internal diameter perpendicular to the long axis of the IVC at the end-expiration, reported in centimeters (cm) from the echocardiogram.
Cardiac Remodeling: Changes in estimated Right Atrial Pressure (RAP) | 6 Months
  This is determined by a combination equation subtracting the venous return (VR) from the central venous pressure (CVP), reported in millimeters of mercury (mmHg) from the echocardiogram.
Cardiac Remodeling: Changes in Right Ventricle Systolic Pressure (RVSP) | 6 Months
  This estimates the pressure inside the artery that supplies the lung with blood, reported in millimeters of mercury (mmHg) from the echocardiogram.
Changes in the rate of mitral annulus velocity (e') | 6 Months
  e' is reported in centimeters per second (cm/s) based on a subject performed echocardiogram
Changes in the ratio of transmitral early peak velocity (E) by pulsed wave Doppler over e' (E/e') | 6 Months
  E/e' is reported as an integer based on the transmitral early peak velocity (E) over the mitral annulus velocity (e') from a subject performed echocardiogram.
PH-HFpEF Only Hemodynamics: Changes in Right Atrial Pressure (RAP) | 6 Months
  This is determined by a combination equation subtracting the venous return (VR) from the central venous pressure (CVP), reported in millimeters of mercury (mmHg) from the echocardiogram.
PH-HFpEF Only Hemodynamics: Changes in Pulmonary Artery Pressure (PAP) | 6 Months
  This is calculated from systolic, by Tricuspid Regurgitation maximum (TRmax) and diastolic, by Pulmonary Regurgitation-end velocity (PR-end) pulmonary artery pressures, reported in millimeters of mercury (mmHg) from the echocardiogram.
PH-HFpEF Only Hemodynamics: Changes in Pulmonary Artery Occlusive Pressure (PAOP) | 6 Months
  This is determined by the pressure value of the pulmonary artery once it's occluded during a Right Heart Catheterization (RHC), measured in millimeters of mercury (mmHg).
PH-HFpEF Only Hemodynamics: Changes in Pulmonary Vascular Resistance (PVR) | 6 Months
  Left Atrial Pressure (LAP), Pulmonary Artery Pressure (PAP) and Cardiac Output (CO) are combined to report the PVR in Wood Units (WU) from a Right Heart Catheterization (RHC).
PH-HFpEF Only Hemodynamics: Changes in Cardiac Output (CO) | 6 Months
  Stoke Volume (SV) and Heart Rate (HR) are combined to report CO in liters per minute (L/min) from the right heart catheterization.
PH-HFpEF Only Hemodynamics: Changes in Cardiac Index (CI) | 6 Months
  Cardiac Output (CO) and Body Surface Area (BSA) are combined to report CI in liters per minute per meters squared (L/min/m^2) from a Right Heart Catherization (RHC).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Jewish Health and University of Colorado Denver, Denver, Colorado
  - Saint Joseph Hospital, Denver, Colorado